CLINICAL TRIAL: NCT01543061
Title: Evaluation of the Effect of Repeated Usage of a New Eyedrop on Silicone Hydrogel Contact Lens Wearers With Dry Eye Complaints
Brief Title: Efficacy Study of a New Eyedrop on Silicone Hydrogel Contact Lens Wearers With Dry Eye Complaints
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Optometric Technology Group Ltd (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AG9965-006 ID 11-19
Record Dates: First submitted 2012-02-22; First posted 2012-03-02 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Contact Lens Related Dry Eye Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- New study eye drop (Active Comparator): One month of contact lens wear with use of the Test study eye drops
  Interventions: Device: OPTIVEtm Plus
- No Eyedrop (Placebo Comparator): One month of contact lens wear with no eye drop use
  Interventions: Procedure: No treatment
- BLINK Contacts Lubricating eye drop (Active Comparator): One month of contact lens wear with use of the Control study eye drops
  Interventions: Device: Blink Contacts® Eye Drops

INTERVENTIONS:
Device: OPTIVEtm Plus — 1 drop in each eye four times a day for a period of 30 (± 3) days
  Arms: New study eye drop
Procedure: No treatment — One month of contact lens wear with no eye drop use
  Arms: No Eyedrop
Device: Blink Contacts® Eye Drops — 1 drop in each eye four times a day for a period of 30 (± 3) days
  Other Names: Blink Contacts®
  Arms: BLINK Contacts Lubricating eye drop

SUMMARY:
The objectives of the investigation will be to assess the effect of the repeated usage of a new eye drop on the tear film characteristics of silicone hydrogel contact lens wearers with contact lens related comfort problems and to quantify any potential benefit.

ELIGIBILITY:
Inclusion criteria:

* Current silicone hydrogel contact lens wearer
* Complaints of contact lens related dry eye (Symptoms and reduced comfortable wearing time)

Exclusion criteria:

* Known allergy or sensitivity to the study product(s) or its components
* Systemic or ocular allergies
* Use of systemic medication which might have ocular side effects.
* Any ocular infection.
* Use of ocular medication.
* Significant ocular tissue anomaly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tear Break up Time | 30 days

SECONDARY OUTCOMES:
Conjunctival staining measurement | 30 days
Tear film evaporation rate | 30 days
Ocular Surface Disease Index questionnaire | 30 days
Comfort, vision and ocular symptoms questionnaire | 30 days
Post wear contact lens deposition and lipid uptake assessment | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michel Guillon, PhD, Principal Investigator — Optometric Technology Group Ltd
Locations (1):
- OTG Research & Consultancy, London, United Kingdom